CLINICAL TRIAL: NCT00355147
Title: Adapting Tools to Implement Stroke Risk Management to Veterans
Acronym: TOOLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IAB 05-297; 0608-01B (Other Grant/Funding Number: US Veterans Health Administration); 1009001684 (Other Grant/Funding Number: US Veterans Health Administration)
Record Dates: First submitted 2006-07-18; First posted 2006-07-21 (Estimated); Results first posted 2015-02-10 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-09

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack
Keywords: Ischemic stroke; Preventive medicine; Transient Ischemic Attack; Neurology; Risk management
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 Secondary Risk Factor Management (Experimental): Patient Secondary Stroke Risk Factor Program including Stroke Self Management and Stroke Peer Support and Physician Stroke Guideline Adherence
  Interventions: Behavioral: Physician stroke guideline adherence; Behavioral: Stroke Self Management
- Attention Control Group (Placebo Comparator): Received Phone Calls from Staff to Control for Attention
  Interventions: Other: Attention Control Group

INTERVENTIONS:
Behavioral: Physician stroke guideline adherence — Provided clinicians with Secondary Stroke Prevention Guidelines/Posted near workstations for Discharge Planning and Provided Clinicians with Seminar on Motivational Interviewing and Goal Setting to Modify Patient Health Behaviors
  Arms: Arm 1 Secondary Risk Factor Management
Behavioral: Stroke Self Management — Provided Post Stroke Guidelines on Secondary Prevention to Clinicians Preparing Discharge Plans; Provided Secondary Stroke Self-Management and Stroke Peer Support to Veteran Patients with Stroke/TIA
  Arms: Arm 1 Secondary Risk Factor Management
Other: Attention Control Group — Received Phone Calls from Staff to Control for Attention
  Arms: Attention Control Group

SUMMARY:
The purpose of this study is to develop and evaluate the local adaptation of existing stroke prevention tools into practice. A stroke prevention program is a collection of materials including written materials like pamphlets and brochures, videotapes and training guides for stroke survivors and evidence based guidelines for the doctors that provide care for them. Other tools that may be used in a stroke prevention program include devices that help patients monitor medical symptoms at home like home blood pressure machines or blood sugar monitors and messaging devices that allow reporting symptoms from home to a health care provider.

We hypothesized Veterans with stroke who receive the Veteran Stroke Prevention Program would engage in better medication compliance and stroke specific quality of life compared to those who did not receive the program.

DETAILED DESCRIPTION:
Stroke affects at least 15,000 veterans each year, and this number will likely increase as the veteran population ages. According to the American Heart Association, the prevalence of stroke is expected to double by 2020 with the increased proportion of older adults nationwide. Our preliminary Quality Enhancement Research Initiative work indicates that stroke risk factors are often undermanaged in the Veterans Health Administration.

This proposed study of a stroke risk factor management program may benefit the Veteran Health System in several ways. First, it offers a systematic program for reduction in stroke risk factors leading to better health for our veterans and a reduction in inpatient and outpatient rehabilitation and home health services for these events. Second, the Veteran Stroke Prevention Program takes into account the varied resources and services offered in VAMCs across the nation, allowing the program to be tailored both to a given facility and to the individual veteran's needs and readiness to change. Importantly, the program could allow all VA facilities to offer guideline-concurrent stroke risk reduction programs and therefore increase compliance with VA/Department of Defense, American Heart Association, and the Joint Commission stroke care guidelines and improve their quality of stroke care.

Comparison(s): We will compare two regionally matched facilities on rates of secondary stroke prevention guideline care during the course of the study at the intervention sites.

ELIGIBILITY:
Inclusion Criteria:

* Veterans 18 years or older hospitalized with stroke or Transient Ischemic Attack at Indianapolis Veterans Administration Medical Center and Houston Veteran Administration Medical Center;
* willing to participate;
* access to telephone;
* speaks and understands English;
* no severe cognitive impairments;
* life expectancy of at least 6 mos;
* willingness to follow-up in Veterans Administration outpatient care.

Exclusion Criteria:

* Severe aphasia or cognitive impairment;
* active alcohol or substance abuse;
* cannot or unwilling to participate;
* does not speak or understand English;
* life expectancy less than 6 mos;
* no access to telephone;
* no Veterans Administration outpatient follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2009-01; Primary Completion 2011-06 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa M. Damush, PhD, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (2):
- United States (2):
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

REFERENCES:
- [Result] Schmid AA, Andersen J, Kent T, Williams LS, Damush TM. Using intervention mapping to develop and adapt a secondary stroke prevention program in Veterans Health Administration medical centers. Implement Sci. 2010 Dec 15;5:97. doi: 10.1186/1748-5908-5-97. PMID 21159171
- [Result] Damush TM, Jackson GL, Powers BJ, Bosworth HB, Cheng E, Anderson J, Guihan M, LaVela S, Rajan S, Plue L. Implementing evidence-based patient self-management programs in the Veterans Health Administration: perspectives on delivery system design considerations. J Gen Intern Med. 2010 Jan;25 Suppl 1(Suppl 1):68-71. doi: 10.1007/s11606-009-1123-5. PMID 20077155
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082
- [Derived] Damush TM, Myers L, Anderson JA, Yu Z, Ofner S, Nicholas G, Kimmel B, Schmid AA, Kent T, Williams LS. The effect of a locally adapted, secondary stroke risk factor self-management program on medication adherence among veterans with stroke/TIA. Transl Behav Med. 2016 Sep;6(3):457-68. doi: 10.1007/s13142-015-0348-6. PMID 27349906

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 Stroke Prevention Intervention: Randomized to receive the intervention which included receipt of stroke prevention and self management intervention and stroke peer support.
- Arm 2 Control Group: Received usual care, follow up telephone calls to control for contact, and educational materials
Period: Overall Study
Arm/Group | Arm 1 Stroke Prevention Intervention | Arm 2 Control Group
Started | 87 | 87
Completed | 69 | 67
Not Completed | 18 | 20
Not completed — Lost to Follow-up | 10 | 8
Not completed — Withdrawal by Subject | 8 | 12

BASELINE CHARACTERISTICS:
Population: Compared groups on strata, age, sex, race/ethnicity, education level, living status, has Caregiver Number of participants were determined by protocol and followed intention to treat. For 3 and 6 month outcomes, we included respondent's last score assuming no change among those with missing data.
Groups:
- Arm 1 Stroke Self Management and Risk Factor Program: Patient Secondary Stroke Risk Factor Program including Stroke Self Management and Stroke Peer Support
  Physician stroke guideline adherence: Provided clinicians with Secondary Stroke Prevention Guidelines/Posted near workstations for Discharge Planning and Provided Clinicians with Seminar on Motivational Interviewing and Goal Setting to Modify Patient Health Behaviors
  Secondary Stroke Self-Management and Risk Factor Management: Provided Post Stroke Guidelines on Secondary Prevention to Clinicians Preparing Discharge Plans; Provided Secondary Stroke Self-Management and Stroke Peer Support to Veteran Patients with Stroke/Transcient Ischemic Attack
- Total: Total of all reporting groups
Arm/Group | Arm 1 Stroke Self Management and Risk Factor Program | Attention Control Group | Total
Number analyzed (Participants) | 87 | 87 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (9.5) | 62.1 (9.4) | 61.3 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Self reported description of respondent's sex
  Participants
    Female | 3 | 2 | 5
    Male | 84 | 85 | 169
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 4 | 15
  Not Hispanic or Latino | 76 | 83 | 159
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 24 | 29 | 53
  White | 54 | 51 | 105
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 7 | 5 | 12
Stroke Specific, Health-Related Quality of Life [Mean (Standard Deviation); unit: units on a scale] — Stroke, specific, health-related quality of life (SSQoL) is a self-reported survey by LS Williams et al Stroke. 1999;30:1362-1369. Includes 12 domains and 49 items which are scored on a 5pt Likert response format with lower score indicating worse function/lower ability on that item or domain. Domain scores were calculated as an unweighted average of item scores in that domain. Overall Total Score was calculated as an unweighted average of domain scores. Each Domain Score and the Overall Total Score all range from 1-5 with 1 being worst and 5 best best.
  units on a scale | 3.72 (0.68) | 3.92 (0.72) | 3.84 (0.72)
Self-Efficacy to Manage Stroke [Mean (Standard Deviation); unit: units on a scale] — This scale is modified from the Arthitis Self-Efficacy scale and is designed to measure Confidence to Manage Stroke Symptoms. The items measure the confidence to manage symptoms and health post stroke on a 1-10 scale where 10 denotes a lot of confidence and a 1 denotes no confidence. The scale score is the average score of the items.
  units on a scale | 7.72 (1.68) | 8.30 (1.60) | 8.14 (1.60)
Self-Efficacy to Communicate with Physician [Mean (Standard Deviation); unit: units on a scale] — The scale designed by K Lorig measures the confidence to communicate with a physician about the patient's health. The response items range from 1-10 where 10 denotes a lot of confidence and a 1 denotes no confidence. The score equals the average of the items.
  units on a scale | 2.08 (0.96) | 2.56 (1.28) | 2.32 (1.16)
Stroke Specific Health Related Quality of Life Perceived Energy [Mean (Standard Deviation); unit: units on a scale] — Perceived Energy Subdomain of the Stroke Specific Quality of Life measures perceived energy after stroke. Item response is on a 5 point Likert scale where 1 denotes worse functioning and 5 denotes best functioning. Domain score was calculated as an unweighted average of item scores in the Energy subdomain.
  units on a scale | 2.62 (1.24) | 3.30 (1.36) | 3.04 (1.36)
Patient Health Questionnaire (PHQ)9 Depressive Symptoms [Mean (Standard Deviation); unit: units on a scale] — PHQ9 is a commonly used scale to measure the degree by which a respondent was bothered by depressive symptoms during the past 2 weeks by Spitzer, Williams, and Kroenke. Each of the 9 items use a 0-3 item response where 0 = "not at all" and 3 ="nearly every day." Total score is the sum of the 9 items.
  units on a scale | 7.72 (6.16) | 6.82 (6.68) | 7.00 (6.34)

OUTCOME MEASURES:

1. Primary Outcome: Stroke Specific Health Related Quality of Life
Description: * Stroke Specifc, Health Related Quality of Life (SSQoL)
  * Self reported survey by LS Williams Weinberger M, Clark, D, Harris L, Biller J. Development of a stroke specific quality of life scale. Stroke, 1999;30:1362-1369.
  * Contains 12 domains and 49 items Scored on a 5 pt Likert response format with lower score indicating worse function/lower ability on that item or domain. Domain scores were calculated as an unweighted average of item scores in that domain. Overall Total Score was calculated as an unweighted average of domain scores.
  We hypothesized the intervention group would report significantly greater stroke specific quality of life than the control group. The level of significance was set to 0.05.
Time Frame: 6 months for (SSQoL) and 3 months for Perceived Energy Subdomain
Population: We hypothesized the intervention group would report significantly greater stroke specific quality of life than the control group. The level of significance was set to 0.05. Number of participants were set per protocol and we used intention to treat in our protocol and analyses. We adjusted the analyses for group, TIA/Stroke, site, and time.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 1 Stroke Self Management and Risk Factor Program: Patient Secondary Stroke Risk Factor Program including Stroke Self Management and Stroke Peer Support
  Physician stroke guideline adherence: Provided clinicians with Secondary Stroke Prevention Guidelines/Posted near workstations for Discharge Planning and Provided Clinicians with Seminar on Motivational Interviewing and Goal Setting to Modify Patient Health Behaviors
  Secondary Stroke Self-Management and Risk Factor Management: Provided Post Stroke Guidelines on Secondary Prevention to Clinicians Preparing Discharge Plans; Provided Secondary Stroke Self-Management and Stroke Peer Support to Veteran Patients with Stroke/TIA
Arm/Group | Arm 1 Stroke Self Management and Risk Factor Program | Attention Control Group
Number analyzed (Participants) | 71 | 68
units on a scale
  Overall Total Score | 3.80 (0.90) | 3.94 (0.82)
  Perceived Energy Score | 2.98 (1.56) | 3.04 (1.42)
Statistical Analysis 1: Comparison: Arm 1 Stroke Self Management and Risk Factor Program vs Attention Control Group; This is an analysis of the outcome, Stroke Specific Quality of Life Overall Total Score; Test type: Superiority or Other; p = 0.69, Mixed Models Analysis; Adjusted for site, strata, baseline score, randomized group, month and the group by month interaction; Mean Difference (Net) = 0.05, Standard Error of Mean 0.11 — This score represents change from baseline to six months across the groups
Statistical Analysis 2: Comparison: Arm 1 Stroke Self Management and Risk Factor Program vs Attention Control Group; This is an analysis of the Perceived Energy Domain within the Stroke Specific Quality of Life Measure; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis — Adjusted for site, strata, baseline value, treatment group, month of assessment, treatment group x month, random subject effect; Mean Difference (Net) = 0.47, Standard Error of Mean 0.23 — This score represents change from baseline to three months across groups

2. Primary Outcome: Self-Efficacy to Manage Stroke Symptoms
Description: Confidence to manage symptoms and health post stroke on a 1-10 scale where 10 denotes a lot of confidence and a 1 denotes no confidence.
Time Frame: 6 months
Population: We hypothesized the intervention group would report significantly greater self-efficacy to manage stroke symptoms than the control group. Level of significance was set to .05. Number of participants were set per protocol and we used intention to treat in our protocol and analyses. We adjusted the analyses for group, TIA/Stroke, site, & time.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 Stroke Self Management and Risk Factor Program | Attention Control Group
Number analyzed (Participants) | 60 | 63
units on a scale | 7.90 (1.78) | 8.08 (1.80)
Statistical Analysis 1: Comparison: Arm 1 Stroke Self Management and Risk Factor Program vs Attention Control Group; Test type: Superiority or Other; p = 0.66, Mixed Models Analysis; Adjusted by site, strata, baseline score, treatment group, month and group by month interaction; Mean Difference (Net) = 0.12 — The score is the change from baseline to six months between groups

3. Secondary Outcome: Medication (Diabetes) Compliance for Secondary Stroke Prevention Risk Factor Managment
Description: * Medication Possession Ratios 6 months post stroke events based upon Pharmacy Refill data
  * Medication Possession Ratios are the % of days in follow up period of 6 months with possession of oral Diabetes drugs (range = 0 -100%)
  * Compliance is defined as Medication Possession Ratio for Diabetes drugs dichotomized as greater than and equal to 80%
Time Frame: baseline, 6 months
Population: We hypothesized the intervention group would report significantly greater medication compliance than the control group. The level of significance was set to 0.05. The number of participants were set per protocol and we used intention to treat in our protocol and analyses.
Measure: Number; unit: participants
Arm/Group | Arm 1 Secondary Risk Factor Management | Attention Control Group
Number analyzed (Participants) | 32 | 14
participants
  >=80% Compliance at baseline | 13 | 8
  <80% Compliance at baseline | 19 | 6
  >=80% Compliance at 6 months | 21 | 6
  <80% Compliance at 6 months | 11 | 8
Statistical Analysis 1: Comparison: Arm 1 Secondary Risk Factor Management vs Attention Control Group; Test type: Superiority or Other; p = 0.06, Regression, Logistic; Odds Ratio (OR) = 6.74, 95% CI 2-sided [0.88 to 51.31]
Statistical Analysis 2: Comparison: Arm 1 Secondary Risk Factor Management; Within group Intervention Pre Post Comparison Compliance with Diabetes Medication; Test type: Superiority or Other; p = 0.036, Regression, Logistic; Odds Ratio (OR) = 3.45, 95% CI 2-sided [1.08 to 10.96]
Statistical Analysis 3: Comparison: Attention Control Group; Within Group attention control group intervention pre post comparison compliance with Diabetes Medication; Test type: Superiority or Other; p = 0.407, Regression, Logistic; Odds Ratio (OR) = 0.51, 95% CI 2-sided [0.10 to 2.70]

4. Secondary Outcome: Medication (Statins) for Secondary Stroke Prevention Risk Factor Management
Description: * Medication Possession Ratios 6 months post stroke event based upon Pharmacy Refill data
  * Medication Possession Ratios are the % of days in follow up period of 6 months with possession of Statin drugs (range= 0-100%).
  * Compliance is defined as Medication Possession Ratio for Statin drugs dichotomized as greater than and equal to 80%.
Time Frame: baseline, 6 months
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Arm 1 Stroke Prevention Intervention | Arm 2 Control Group
Number analyzed (Participants) | 72 | 71
participants
  >=80% Compliance at baseline | 16 | 18
  <80% Compliance at baseline | 56 | 53
  >=80% Compliance at 6 months | 44 | 39
  <80% Compliance at 6 months | 28 | 32
Statistical Analysis 1: Comparison: Arm 1 Stroke Prevention Intervention vs Arm 2 Control Group; Between Group Intervention Pre Post Comparison Compliance with Statin Medication; Test type: Superiority or Other; p = 0.05, Regression, Logistic; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.54 to 4.48]
Statistical Analysis 2: Comparison: Arm 1 Stroke Prevention Intervention; Within Group Intervention Pre Post Comparison Compliance with Statin Medication; Test type: Superiority or Other; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 5.98, 95% CI 2-sided [2.81 to 12.76]
Statistical Analysis 3: Comparison: Arm 2 Control Group; Within Group Attention Control Pre Post Comparison Compliance with Statin Medication; Test type: Superiority or Other; p = 0.0004, Regression, Logistic; Odds Ratio (OR) = 3.83, 95% CI 2-sided [1.83 to 8.01]

5. Secondary Outcome: Medication (Hypertension) Compliance for Secondary Stroke Prevention Risk Factor Management
Description: * Medication Possession Ratios 6 months post stroke event based upon Pharmacy Refill data
  * Medication Possession Ratios are the % of days in follow up period of 6 months with possession of hypertension drugs (range = 0-100%)
  * Compliance is defined as Medication Possession Ratio for Hypertension drugs dichotomized as greater than and equal to 80%.
Time Frame: Baseline, 6 months
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Arm 1 Stroke Self Management and Risk Factor Program | Attention Control Group
Number analyzed (Participants) | 79 | 70
participants
  >=80% Compliance at baseline | 39 | 41
  <80% Compliance at baseline | 40 | 29
  >=80% Compliance at 6 months | 61 | 48
  <80% Compliance at 6 months | 18 | 22
Statistical Analysis 1: Comparison: Arm 1 Stroke Self Management and Risk Factor Program vs Attention Control Group; Between Group Intervention Pre Post Comparison Compliance with Hypertension Medication; Test type: Superiority or Other; p = 0.096, Regression, Logistic; Odds Ratio (OR) = 2.34, 95% CI 2-sided [0.86 to 6.40]
Statistical Analysis 2: Comparison: Arm 1 Stroke Self Management and Risk Factor Program; Within Group Intervention Pre Post Comparison Compliance with Hypertension Medication; Test type: Superiority or Other; p = 0.0004, Regression, Logistic; Odds Ratio (OR) = 3.68, 95% CI 2-sided [1.81 to 7.48]
Statistical Analysis 3: Comparison: Attention Control Group; Within Group Attention Group Pre Post Comparison Compliance with Hypertension Medication; Test type: Superiority or Other; p = 0.21, Regression, Logistic; Odds Ratio (OR) = 1.57, 95% CI 2-sided [0.77 to 3.21]

ADVERSE EVENTS:
Time Frame: Continuously throughout study intervention period of 6 months
Arm/Group | Arm 1 Stroke Self Management and Risk Factor Program | Attention Control Group
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/87
Other Adverse Events (participants affected / at risk) | 0/87 | 0/87

LIMITATIONS AND CAVEATS:
Both our intervention and control groups experienced attrition during the study period but the rate between groups did not differ significantly.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes